CLINICAL TRIAL: NCT01848353
Title: Incentivizing Behavior: Promoting More Physical Activity in American Indian Youth
Brief Title: Financial Incentives to Exercise for Adolescents
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P20 MD000528-RP2; P20MD000528 (NIH)
Record Dates: First submitted 2013-04-25; First posted 2013-05-07 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Insulin Resistance; Obesity; Sedentary Lifestyle
MeSH Terms: conditions — Insulin Resistance; Obesity; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Standard payment, phase 1 (Active Comparator): All participants will perform exercise training. Participants in this arm will receive a fixed amount of money for exercise session lasting at least 20 minutes during weeks 1-16 (phase 1). All exercise recommendations and outcome tests will be same for this group as the experimental group so that the two groups differ only in the financial incentives they receive for exercise behavior.
  Interventions: Behavioral: Exercise training
- Standard payment, phase 2 (Active Comparator): All participants will perform exercise training. Participants in this arm will receive a fixed amount of money for exercise session lasting at least 20 minutes during weeks 17-32 (phase 2). All exercise recommendations and outcome tests will be same for this group as the experimental group so that the two groups differ only in the financial incentives they receive for exercise behavior.
  Interventions: Behavioral: Exercise training
- Ramp-down payment, phase 3 (Active Comparator): All participants will perform exercise training. This phase will last from weeks 33-48 (phase 3). Participants in this arm will receive a fixed amount of money for exercise session lasting at least 20 minutes, but the value of the payments will decrease weekly (ramp-down) until reaching zero in week 41. All exercise recommendations and outcome tests will be same for this group as the experimental group so that the two groups differ only in the financial incentives they receive for exercise behavior.
  Interventions: Behavioral: Exercise training
- Incentivized payment, phase 1 (Experimental): All participants will perform exercise training. Participants in this arm will receive an increasing amount of money when they increase exercise frequency (number of days) during weeks 1-16 (phase 1). All exercise recommendations and outcome tests will be same for this group as the active comparator group so that the two groups differ only in the financial incentives they receive for exercise behavior
  Interventions: Behavioral: Exercise training
- Incentivized payment, phase 2 (Experimental): All participants will perform exercise training. Participants in this arm will receive an increasing amount of money when they exercise for longer than 20 minutes per session during weeks 17-32 (phase 2). All exercise recommendations and outcome tests will be same for this group as the active comparator group so that the two groups differ only in the financial incentives they receive for exercise behavior
  Interventions: Behavioral: Exercise training
- Raffle payment, phase 3 (Experimental): All participants will perform exercise training. In weeks 33-48 (phase 3)participants in this arm will receive fewer financial incentives than in the prior 32 weeks but they will be delivered through a raffle system to utilize a variable reinforcement approach. All exercise recommendations and outcome tests will be same for this group as the active comparator group so that the two groups differ only in the financial incentives they receive for exercise behavior.
  Interventions: Behavioral: Exercise training
- Normal weight, low activity group (No Intervention): This group of participants will complete only the baseline tests and assessments and will serve as a reference group. They will be selected to have low physical activity and fitness like the intervention group. Therefore differences in their results with the intervention group will reflect the effects of overweight/obesity on the variables of interest.
- Normal weight, high activity group (No Intervention): This group of participants will complete only the baseline tests and assessments and will serve as a reference group. They will be selected to have higher physical activity and fitness than the intervention group. They will therefore serve as a healthy reference group and differences in their results with the intervention group will reflect the effects of both overweight/obesity and physical activity on the variables of interest.

INTERVENTIONS:
Behavioral: Exercise training — All participants will perform exercise training at the wellness center. Exercise duration and intensity will be recorded with heart rate monitors.
  Arms: Incentivized payment, phase 1; Incentivized payment, phase 2; Raffle payment, phase 3; Ramp-down payment, phase 3; Standard payment, phase 1; Standard payment, phase 2

SUMMARY:
Among youth populations, American Indians have the highest prevalence of diabetes in the United States. This study will use exercise as the principal lifestyle modification approach to reduce the risk of diabetes in this population. The Choctaw Nation of Oklahoma has several excellent, but underutilized wellness facilities in their Health Services Area in rural Southeast Oklahoma, a low socioeconomic region. It has been established that exercise lowers diabetes risk, and many overweight/obese, insulin resistant American Indian youth who live in this region would benefit from an increase in regular exercise. The challenge is to modify behavior so that routine exercise is established and maintained. The proposed study will test whether monetary incentives can elicit greater frequency and duration of exercise in American Indian youth when transportation and access barriers are reduced.

DETAILED DESCRIPTION:
Study participants in the intervention arm of the study will be asked to exercise on 3 days per week for 48 weeks. Clinical and physical assessments will be performed at baseline and after 16, 32 and 48 weeks. Participants will be randomized into one of two groups. Each group will receive payment for exercise sessions completed but one group will be on a fixed schedule of compensation and the other will have a schedule that incentivizes frequency or duration of exercise. In addition, two reference groups of age-matched participants who are normal weight and subclassified as having either low or high levels of physical activity and fitness will be tested. The reference groups will complete baseline tests and will not enter the exercise intervention program.

ELIGIBILITY:
Inclusion Criteria for exercise intervention cohort:

* 11.0-20.9 years old
* overweight or obese
* family history of diabetes (primary or secondary relative)
* not in sports or exercise program (3 or fewer days per week of moderate-to-vigorous intensity physical activity, MVPA) for prior 3 months
* Tanner stage 2 or above

Inclusion Criteria for reference group cohort:

* 11.0-20.9 years old
* normal weight
* For low physical activity subgroup: not in sports or exercise program (3 or fewer days per week of MVPA) for prior 3 months
* For high physical activity subgroup: >30 minutes of structured MVPA on >3 days/week over the preceding 3 months
* Tanner stage 2 or above

Exclusion Criteria for all participants:

* metabolic, endocrine, cardiovascular, kidney disease
* orthopedic problems that limit physical activity
* medications or treatments that would interfere with the outcomes and interpretations
* smoking or tobacco use
* alcohol or illicit drug use
* pregnancy

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 142 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Short, PhD, Principal Investigator — University of Oklahoma; Kenneth C Copeland, MD, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - Choctaw Nation of Oklahoma Healthcare, Hugo, Oklahoma
  - Choctaw Nation Diabetes Wellness Center, Talihina, Oklahoma

REFERENCES:
- [Derived] Short KR, Chadwick JQ, Cannady TK, Branam DE, Wharton DF, Tullier MA, Thompson DM, Copeland KC. Using financial incentives to promote physical activity in American Indian adolescents: A randomized controlled trial. PLoS One. 2018 Jun 1;13(6):e0198390. doi: 10.1371/journal.pone.0198390. eCollection 2018. PMID 29856832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the exercise intervention was July 2013 - April 2016. Recruitment for the reference group was July 2015 - April 2017. All participants were were recruited from medical clinics, schools, or community settings in Southeast Oklahoma.
Pre-assignment Details: 142 people enrolled (completed informed consent). During screening, 4 OW/Ob and 8 NW people were disqualified, and 5 OW/Ob and 5 NW people voluntarily withdrew. Baseline data were thus available for 120 people. After baseline testing was complete, 81 OW/Ob participants were randomly assigned to either standard pay or incentive group for Phase 1.
Groups:
- Standard Payment: All participants will perform exercise training. Participants in this arm will receive a fixed amount of money for exercise session lasting at least 20 minutes. All exercise recommendations and outcome tests will be same for this group as the experimental group so that the two groups differ only in the financial incentives they receive for exercise behavior.
  Exercise training: All participants will perform exercise training at the wellness center. Exercise duration and intensity will be recorded with heart rate monitors.
- Incentivized Payment: All participants will perform exercise training. Participants in this arm will receive an increasing amount of money when they increase exercise frequency (number of days) during weeks 1-16 (phase 1), or increase exercise duration (minutes per session) during weeks 17-32 (phase 2). In phase 3 the payment will be a lottery, with the number of lottery chances based on exercise frequency and duration. All exercise recommendations and outcome tests will be same for this group as the active comparator group so that the two groups differ only in the financial incentives they receive for exercise behavior
  Exercise training: All participants will perform exercise training at the wellness center. Exercise duration and intensity will be recorded with heart rate monitors.
Period: Phase 1
Arm/Group | Standard Payment | Incentivized Payment | Normal Weight, Low Activity Group | Normal Weight, High Activity Group
Started | 38 | 43 | 20 | 19
Completed | 35 | 42 | 20 | 19
Not Completed | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Period: Phase 2
Arm/Group | Standard Payment | Incentivized Payment | Normal Weight, Low Activity Group | Normal Weight, High Activity Group
Started | 23 (26 participants from Phase 1 intervention (both groups) withdrew and did not complete Phase 2) | 28 (26 participants from Phase 1 intervention (both groups) withdrew and did not complete Phase 2) | 0 (Normal weight participants only completed baseline testing in Phase 1.) | 0 (Normal weight participants only completed baseline testing in Phase 1.)
Completed | 20 | 26 | 0 | 0
Not Completed | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 0
Period: Phase 3
Arm/Group | Standard Payment | Incentivized Payment | Normal Weight, Low Activity Group | Normal Weight, High Activity Group
Started | 5 (31 participants from Phase 2 intervention (both groups) withdrew and did not complete Phase 3) | 10 (31 participants from Phase 2 intervention (both groups) withdrew and did not complete Phase 3) | 0 (Normal weight participants only completed baseline testing in Phase 1.) | 0 (Normal weight participants only completed baseline testing in Phase 1.)
Completed | 4 | 9 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Normal weight groups completed only the baseline testing. The overweight/obese group entered the exercise program at phase 1, and then continued on to phases 2 and 3 if they remained enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Payment, Phase 1 | Incentivized Payment, Phase 1 | Normal Weight, Low Activity Group | Normal Weight, High Activity Group | Total
Number analyzed (Participants) | 38 | 43 | 20 | 19 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (2.2) | 14.2 (2.2) | 14.6 (2.3) | 14.3 (1.9) | 14.4 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 11 | 7 | 64
  Male | 17 | 18 | 9 | 12 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 38 | 43 | 20 | 19 | 120
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 43 | 20 | 19 | 186
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 33.4 (7.0) | 34.8 (6.1) | 20.8 (1.9) | 20.1 (2.4) | 30.1 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Volume of Exercise (Total Time)
Description: Frequency and duration of moderate-to-vigorous physical activity will be measured using heart rate monitors. The monitors will be worn each exercise session. Participants are asked to complete 3 exercise sessions per week throughout the 48-week period of enrollment. The primary comparison between the experimental and active comparator groups will be the volume of exercise (total time) accumulated. Comparisons will be made for accumulated exercise volume at 16, 32, and 48 weeks and the change from baseline (week 0).
Time Frame: at baseline (week 0) and weeks 16, 32, and 48.
Population: In Phase 1, 81 people were randomized, but 4 withdrew after assignment so 77 people had exercise behavior data for analyses. In Phase 2, 51 were randomized, but 5 withdrew after assignment, leaving 46 for behavior analyses. In Phase 3, 15 were randomized, 2 withdrew after assignment, leaving 13 for behavior analyses.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard Payment, Phase 1 | Incentivized Payment, Phase 1 | Standard Payment, Phase 2 | Incentivized Payment, Phase 2 | Ramp-down Payment, Phase 3 | Raffle Payment, Phase 3
Number analyzed (Participants) | 35 | 42 | 20 | 26 | 4 | 9
hours | 15.2 (10.1) | 15.0 (8.1) | 8.0 (5.5) | 12.4 (11.1) | 10.2 (3.8) | 8.8 (4.7)

2. Secondary Outcome: Insulin Resistance
Description: Fasting blood glucose and insulin concentration will be measured and used to calculate the homeostatic model of assessment for insulin resistance (iHOMA2, %S). Testing will be performed at baseline (week 0) and weeks 16, 32, and 48. Data analysis will focus on the change from baseline and whether that change differs between groups.
Time Frame: at baseline (week 0) and weeks 16, 32, and 48.
Population: In Phase 1, 20 out of 77 people who started were lost to follow-up so post-test data were not available. In Phase 2, 26 out of 46 people who started were lost to follow-up. In Phase 3, 3 out of 13 people who started were lost to follow-up.
Measure: Mean (Standard Deviation); unit: % of sensitivity
Arm/Group | Standard Payment, Phase 1 | Incentivized Payment, Phase 1 | Standard Payment, Phase 2 | Incentivized Payment, Phase 2 | Ramp-down Payment, Phase 3 | Raffle Payment, Phase 3 | Normal Weight, Low Activity Group | Normal Weight, High Activity Group
Number analyzed (Participants) | 25 | 32 | 9 | 11 | 4 | 6 | 20 | 19
% of sensitivity | 75 (49) | 69 (44) | 66 (36) | 77 (45) | 57 (28) | 65 (35) | 170 (75) | 179 (92)

3. Secondary Outcome: Exercise Fitness
Description: Peak oxygen uptake (VO2max) during a progressive intensity bicycle test to fatigue. Testing will be performed at baseline (week 0) and weeks 16, 32, and 48. Data analysis will focus on the change from baseline and whether that change differs between groups.
Time Frame: at baseline (week 0) and weeks 16, 32, and 48.
Population: In Phase 1, 20 out of 77 people who started were lost to follow-up so post-test data were not available. In Phase 2, 26 out of 46 people who started were lost to follow-up. In Phase 3, 3 out of 13 people who started were lost to follow-up. Missing data: 2 people in Phase 1 (1 in each group), 1 person in NW low activity group.
Measure: Mean (Standard Deviation); unit: ml/kg fat free mass/minute
Arm/Group | Standard Payment, Phase 1 | Incentivized Payment, Phase 1 | Standard Payment, Phase 2 | Incentivized Payment, Phase 2 | Ramp-down Payment, Phase 3 | Raffle Payment, Phase 3 | Normal Weight, Low Activity Group | Normal Weight, High Activity Group
Number analyzed (Participants) | 24 | 31 | 9 | 11 | 4 | 6 | 19 | 19
ml/kg fat free mass/minute | 36.9 (8.0) | 37.4 (8.6) | 39.0 (10.8) | 39.2 (12.9) | 39.2 (5.8) | 43.0 (6.6) | 61.7 (7.5) | 45.1 (5.4)

4. Secondary Outcome: Body Composition
Description: Body fat content. Testing will be performed at baseline (week 0) and weeks 16, 32, and 48. Data analysis will focus on the change from baseline and whether that change differs between groups.
Time Frame: at baseline (week 0) and weeks 16, 32, and 48.
Population: In Phase 1, 20 out of 77 people who started were lost to follow-up so post-test data were not available. In Phase 2, 26 out of 46 people who started were lost to follow-up. In Phase 3, 3 out of 13 people who started were lost to follow-up. Missing data: 1 person in NW Lo fit group.
Measure: Mean (Standard Deviation); unit: Total body fat percentage
Arm/Group | Standard Payment, Phase 1 | Incentivized Payment, Phase 1 | Standard Payment, Phase 2 | Incentivized Payment, Phase 2 | Ramp-down Payment, Phase 3 | Raffle Payment, Phase 3 | Normal Weight, Low Activity Group | Normal Weight, High Activity Group
Number analyzed (Participants) | 25 | 32 | 9 | 11 | 4 | 6 | 19 | 19
Total body fat percentage | 43.9 (7.8) | 44.4 (7.7) | 40.8 (4.4) | 40.9 (7.1) | 40.4 (3.5) | 44.9 (9.1) | 21.2 (6.3) | 23.3 (7.7)

5. Other Pre Specified Outcome: Physical Activity
Description: Daily step counts measured with accelerometers. Testing will be performed at baseline (week 0) and weeks 16, 32, and 48. Data analysis will focus on the change from baseline and whether that change differs between groups.
Time Frame: at baseline (week 0) and weeks 16, 32, and 48.
Population: In Phase 1, 20 of 77 starters lost to follow-up (no post-test data). In Phase 2, 26 of 46 starters lost to follow-up. In Phase 3, 3 of 13 starters lost to follow-up. Missing data: Phase 1 (4 std, 5 incentive), Phase 2 (2 std, 3 incentive), Phase 3 (1 std, 2 incentive), NW (1 Low, 1 High).
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Standard Payment, Phase 1 | Incentivized Payment, Phase 1 | Standard Payment, Phase 2 | Incentivized Payment, Phase 2 | Ramp-down Payment, Phase 3 | Raffle Payment, Phase 3 | Normal Weight, Low Activity Group | Normal Weight, High Activity Group
Number analyzed (Participants) | 21 | 27 | 7 | 8 | 3 | 4 | 19 | 18
steps per day | 6048 (2711) | 6028 (3136) | 4862 (1217) | 6787 (4273) | 4166 (1882) | 6863 (2321) | 9492 (3176) | 8338 (3103)

6. Other Pre Specified Outcome: Blood Lipids
Description: Standard assessment of fasting triglycerides. Testing will be performed at baseline (week 0) and weeks 16, 32, and 48. Data analysis will focus on the change from baseline and whether that change differs between groups.
Time Frame: at baseline (week 0) and weeks 16, 32, and 48.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Standard Payment, Phase 1 | Incentivized Payment, Phase 1 | Standard Payment, Phase 2 | Incentivized Payment, Phase 2 | Ramp-down Payment, Phase 3 | Raffle Payment, Phase 3 | Normal Weight, Low Activity Group | Normal Weight, High Activity Group
Number analyzed (Participants) | 25 | 32 | 9 | 11 | 4 | 6 | 20 | 19
mg/dl | 92 (56) | 97 (68) | 64 (30) | 114 (87) | 83 (50) | 102 (80) | 51 (24) | 60 (30)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each participant for as long as they were actively enrolled in the study, a period of up to 48 weeks for the exercise intervention group.
Description: Injury or illness due to exercise performed as part of the study
Arm/Group | Standard Payment, Phase 1 | Incentivized Payment, Phase 1 | Standard Payment, Phase 2 | Incentivized Payment, Phase 2 | Ramp-down Payment, Phase 3 | Raffle Payment, Phase 3 | Normal Weight, Low Activity Group | Normal Weight, High Activity Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/43 | 0/23 | 0/28 | 0/5 | 0/10 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/43 | 0/23 | 0/28 | 0/5 | 0/10 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/38 | 0/43 | 0/23 | 0/28 | 0/5 | 0/10 | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT01848353/Prot_SAP_000.pdf